CLINICAL TRIAL: NCT04992390
Title: A Randomised Optimisation Study of a Brief Digital Imagery-competing Task Intervention to Support NHS ICU Staff Experiencing Intrusive Memories of Traumatic Events From Working in the COVID-19 Pandemic
Brief Title: A Brief GAmeplay Intervention for NHS ICU Staff Affected by COVID-19 Trauma (GAINS Study)
Acronym: GAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P1vital Products Limited (Industry)
Collaborators: Wellcome Trust (Other); Uppsala University (Other); Intensive Care Society (Unknown); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P1V-GAINS-IN01
Record Dates: First submitted 2021-08-02; First posted 2021-08-05 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Intrusive Memories of Traumatic Event(s)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention arm (Experimental): Immediate access to the brief digital imagery-competing task intervention plus symptom monitoring for 4 weeks including completing a daily count of the number of their intrusive memories in week 4 (primary outcome).
  Interventions: Behavioral: Brief digital imagery-competing task intervention
- Delayed intervention arm (Experimental): Usual care for 4 weeks including completing a daily count of the number of their intrusive memories in week 4 (primary outcome), followed by access to the brief digital imagery-competing task intervention plus symptom monitoring for 4 weeks.
  Interventions: Behavioral: Brief digital imagery-competing task intervention

INTERVENTIONS:
Behavioral: Brief digital imagery-competing task intervention — First session guided by a researcher: A memory cue followed by playing the brief digital imagery-competing task with mental rotation instructions.
  Option to engage in self-administered/guided sessions after the first session and record their intrusive memories (symptom monitoring).

SUMMARY:
Intensive care unit (ICU) staff are frequently exposed to traumatic events at work (e.g., witnessing patients die), amplified by the COVID-19 pandemic. A significant proportion experience intrusive memories of these events that pop suddenly into mind: these imagery-based memories can disrupt functioning and contribute to posttraumatic stress disorder. Previous research has shown that a brief behavioural intervention can reduce the number of intrusive memories after a traumatic event. In this study we aim to optimise a brief digital intervention to help reduce the number of intrusive memories experienced by ICU staff (primary outcome). We will explore if it can improve work functioning and wellbeing (secondary outcomes). We will recruit approximately 150 ICU staff with intrusive memories of events experienced during the COVID-19 pandemic.

The study is funded by the Wellcome Trust (223016/Z/21/Z).

DETAILED DESCRIPTION:
A statistical analysis plan was prepared prior to the first interim analysis for the outcomes that guided study optimisation, i.e., primarily the primary outcome.

A second statistical analysis plan was prepared prior to the end of the study, outlining the standard (frequentist) statistical approaches used to analyse the primary, secondary and tertiary data.

Regular monitoring performed by P1vital Products to verify that the study is conducted and data are generated, documented and reported in compliance with the protocol, GCP and the applicable regulatory requirements.

Quality assurance representatives from the Sponsor may carry out an audit of the study in compliance with regulatory guidelines and relevant standard operating procedures.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 or above.
* Able to read, write and speak in English.
* Worked in a clinical role in an NHS Intensive Care Unit or equivalent during the COVID-19 pandemic (e.g. as a member of ICU staff or deployed to work in the ICU during the pandemic)
* Experienced at least one traumatic event related to their work during the COVID-19 pandemic, meeting criterion A of the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for Post-Traumatic Stress Disorder (PTSD): "exposure to actual or threatened death, serious injury, or sexual violence" by "directly experiencing the traumatic event(s)" or "witnessing, in person, the event(s) as it occurred to others"
* Experience intrusive memories of the traumatic event(s).
* Experienced at least three intrusive memories in the week prior to screening.
* Have internet access.
* Willing and able to provide informed consent and complete study procedures (including briefly listing their intrusive memories (without going into any detail), and playing the brief digital imagery-competing task with particular mental rotation instructions, and completing an online intrusive memory diary).
* Willing and able to be contacted by the research team during the study period.

Exclusion criteria:

• Have fewer than three intrusive memories during the run-in week.

We will not exclude those undergoing other treatment for PTSD or its symptoms, so the study is as inclusive as possible to meet the challenges ICU staff are facing during the COVID-19 pandemic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Principal Investigator — Uppsala University
Locations (1):
- P1vital Products Limited, Wallingford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised database of individual participant data, along with a data dictionary, as well as the Clinical Study Report (which will include summarised anonymised participant data), will be shared on the Open Science Framework.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Study Protocol and Statistical Analysis Plan were made available on the Open Science Framework prior to LPLV. An executive summary of the Clinical Study Report was shared following publication. These together with supporting information (see below) are available indefinitely and with no end date on Open Science Framework Platform.
Access Criteria: Anonymised research data will be made available on open science frame work (OSF) indefinitely.
  OSF is an open source web application that is freely accessible to public and scientific community.
  OSF links are:
  Protocol, Optimisation SAP (Bayesian) and Descriptive SAP (Frequentist):
  https://osf.io/2xn5m/
  Bayesian paper analysis scripts, database and data code book:
  https://osf.io/m5cvj/
  Frequentist paper analysis scripts, database and data code book: https://osf.io/j9v2z/
URL: https://osf.io/2xn5m/

REFERENCES:
- [Background] Iyadurai L, Highfield J, Kanstrup M, Markham A, Ramineni V, Guo B, Jaki T, Kingslake J, Goodwin GM, Summers C, Bonsall MB, Holmes EA. Reducing intrusive memories after trauma via an imagery-competing task intervention in COVID-19 intensive care staff: a randomised controlled trial. Transl Psychiatry. 2023 Sep 1;13(1):290. doi: 10.1038/s41398-023-02578-0. PMID 37658043
- [Result] Ramineni V, Millroth P, Iyadurai L, Jaki T, Kingslake J, Highfield J, Summers C, Bonsall MB, Holmes EA. Treating intrusive memories after trauma in healthcare workers: a Bayesian adaptive randomised trial developing an imagery-competing task intervention. Mol Psychiatry. 2023 Jul;28(7):2985-2994. doi: 10.1038/s41380-023-02062-7. Epub 2023 Apr 26. PMID 37100869
- See also: Published paper of primary outcome results (Bayesian analysis) — https://www.nature.com/articles/s41380-023-02062-7
- See also: Published paper of primary outcome results (Frequentist analysis) — https://pubmed.ncbi.nlm.nih.gov/37658043/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 106 Participants provided informed consent to participate. 4 participants did not meeting inclusion criteria after which 102 commenced run-in week intrusive memory diary.
  88 participants were eligible after run-in week. 1 participant became lost to follow-up and 1 participant withdrew.
  86 Participants were randomised (n=43 immediate arm; n=43 delayed arm).
Groups:
- Immediate Intervention Arm: Immediate access to the brief digital imagery-competing task intervention plus symptom monitoring for 4 weeks including completing a daily count of the number of their intrusive memories in week 4 (primary outcome).
  Brief digital imagery-competing task intervention: First session guided by a researcher: A memory cue followed by playing the brief digital imagery-competing task with mental rotation instructions.
  Option to engage in self-administered/guided sessions after the first session and record their intrusive memories (symptom monitoring).
- Delayed Intervention Arm: Usual care for 4 weeks including completing a daily count of the number of their intrusive memories in week 4 (primary outcome), followed by access to the brief digital imagery-competing task intervention plus symptom monitoring for 4 weeks.
  Brief digital imagery-competing task intervention: First session guided by a researcher: A memory cue followed by playing the brief digital imagery-competing task with mental rotation instructions.
  Option to engage in self-administered/guided sessions after the first session and record their intrusive memories (symptom monitoring).
- Participants Who Commenced run-in Week But Were Not Randomised.: This study used a run-in week to establish a baseline number of intrusive memories over a seven-day period.
  Participants were randomised if they completed the run-in week and recorded at least three intrusive memories during the run-in week, and completed baseline questionnaires. As such, not all participants who commenced the run-in week completed baseline questionnaire and thus could not be randomised to either the immediate or delayed intervention arms.
  No data are available for those participants were not randomised.
Period: Run-In/Screening Week
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 43 | 43 | 16
Completed | 43 | 43 | 2
Not Completed | 0 | 0 | 14
Not completed — Recorded fewer than three intrusive memories | 0 | 0 | 7
Not completed — Lost to Follow-up | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Baseline Questionnaires
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 43 | 43 | 2
Completed | 43 | 43 | 0
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Immediate Arm Receive Intervention
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 43 | 43 | 0
Completed (Only participants in the Immediate Intervention Arm received their allocated intervention at this stage. Those in the Delayed Intervention Arm received the allocated intervention after crossover.) | 40 | 43 | 0
Not Completed | 3 | 0 | 0
Period: Week 4 Primary Outcome
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 40 | 43 | 0
Completed | 36 | 39 | 0
Not Completed | 4 | 4 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Did not complete week 4 diary but not lost to follow-up | 1 | 0 | 0
Period: Week 4 Secondary Outcomes
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 37 (Please note, the non-completion of prior outcome measures did not prevent participants from progressing to later stages of the study.) | 39 | 0
Completed | 28 | 38 | 0
Not Completed | 9 | 1 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Secondary questionnaires missing/partially complete | 5 | 1 | 0
Period: Delayed Arm Receive Intervention
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 33 (Please note, the non-completion of prior outcome measures did not prevent participants from progressing to later stages of the study.) | 39 (Please note, the non-completion of prior outcome measures did not prevent participants from progressing to later stages of the study.) | 0
Completed (Only participants in the Delayed Intervention Arm received their allocated intervention at this stage (after crossover).) | 33 | 38 | 0
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Week 8 Replication After Crossover
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started (In week 8, the intrusive memory daily diary was completed ONLY by the delayed arm.) | 33 | 38 | 0
Completed | 33 | 32 | 0
Not Completed | 0 | 6 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Week 8 - Other Secondary Outcomes
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Participants Who Commenced run-in Week But Were Not Randomised.
Started | 33 | 32 | 0
Completed | 31 | 29 | 0
Not Completed | 2 | 3 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Secondary questionnaires partially complete | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomised to an intervention condition (groups combined, n=86)
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.8) | 39.9 (9.9) | 38.7 (9.9)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Participants
    Gender: number analyzed (Participants) | 42 | 42 | 84
    Gender: Woman | 34 | 35 | 69
    Gender: Man | 8 | 7 | 15
    Gender: Other (Transwoman; Transman; Gender-variant/non-binary; Other Identity; Prefer not to answer) | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Participants
    Ethnicity: number analyzed (Participants) | 42 | 42 | 84
    Ethnicity: White - British | 18 | 18 | 36
    Ethnicity: White - Irish | 1 | 1 | 2
    Ethnicity: White - Any other White background | 9 | 14 | 23
    Ethnicity: Mixed - Any other mixed background | 2 | 0 | 2
    Ethnicity: Asian - Indian | 2 | 3 | 5
    Ethnicity: Asian - Any other Asian background | 1 | 0 | 1
    Ethnicity: Black - African | 1 | 1 | 2
    Ethnicity: Other - Any other ethnic group | 0 | 1 | 1
    Ethnicity: Unknown - Not stated | 8 | 4 | 12
    Ethnicity: Other categories (see publication for specification of other categories) | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Participants
    number analyzed (Participants) | 42 | 42 | 84
    Single | 13 | 13 | 26
    Living apart from partner | 1 | 0 | 1
    Married or cohabiting | 25 | 28 | 53
    Divorced or separated | 3 | 1 | 4
    Other categories (Widowed; Other) | 0 | 0 | 0
Work and Employment, Number of hours worked per week [Mean (Standard Deviation); unit: Hours (per week)] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Hours (per week)
    number analyzed (Participants) | 42 | 42 | 84
    (all) | 37.9 (13.3) | 37.8 (9.2) | 37.8 (11.4)
Work and Employment, Time as healthcare professional (years) [Mean (Standard Deviation); unit: Years] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Years
    number analyzed (Participants) | 42 | 42 | 84
    (all) | 13.0 (8.6) | 16.4 (10.8) | 14.7 (9.8)
Employment Status [Count of Participants; unit: Participants] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Participants
    number analyzed (Participants) | 42 | 42 | 84
    Working full time | 34 | 32 | 66
    Working part time | 6 | 10 | 16
    Sick leave | 1 | 0 | 1
    Other | 1 | 0 | 1
    Other categories (Jobseeking; Student; Retired) | 0 | 0 | 0
NHS Job Role [Count of Participants; unit: Participants]
  Allied Health Professionals | 3 | 1 | 4
  Doctors | 8 | 11 | 19
  Health Informatics | 0 | 1 | 1
  Healthcare Support Worker | 2 | 1 | 3
  Nursing | 29 | 28 | 57
  Other/unknown | 0 | 1 | 1
  Pharmacy | 1 | 0 | 1
Health Background [Count of Participants; unit: Participants] — Population: Total n observed for data is 83 (delayed arm n=42; immediate arm n=41)
  Participants
    Do you have any current physical health problems e.g. diabetes, heart problems?: number analyzed (Participants) | 41 | 42 | 83
    Do you have any current physical health problems e.g. diabetes, heart problems?: Yes | 8 | 9 | 17
    Do you have any current physical health problems e.g. diabetes, heart problems?: No | 33 | 33 | 66
    Have you been treated for/diagnosed with any mental health problems e.g. depression, anxiety, PTSD?: number analyzed (Participants) | 41 | 42 | 83
    Have you been treated for/diagnosed with any mental health problems e.g. depression, anxiety, PTSD?: Yes | 22 | 24 | 46
    Have you been treated for/diagnosed with any mental health problems e.g. depression, anxiety, PTSD?: No | 19 | 18 | 37
    Are you receiving any current treatments/medications for these?: number analyzed (Participants) | 41 | 42 | 83
    Are you receiving any current treatments/medications for these?: Yes | 15 | 17 | 32
    Are you receiving any current treatments/medications for these?: No | 26 | 25 | 51
    Has anyone in your close family been treated for/diagnosed with any mental health problems?: number analyzed (Participants) | 41 | 42 | 83
    Has anyone in your close family been treated for/diagnosed with any mental health problems?: Yes | 14 | 16 | 30
    Has anyone in your close family been treated for/diagnosed with any mental health problems?: No | 27 | 26 | 53
Experiences of Prior Trauma [Mean (Standard Deviation); unit: Number of events experienced/witnessed] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42)
  Number of events experienced/witnessed
    How many work-related traumatic events have you experienced/witnessed during COVID-19?: number analyzed (Participants) | 42 | 42 | 84
    How many work-related traumatic events have you experienced/witnessed during COVID-19? | 35.9 (58.0) | 38.4 (80.9) | 37.1 (70.0)
    How many traumatic events that were not work-related have you experienced/witnessed during COVID-19?: number analyzed (Participants) | 42 | 42 | 84
    How many traumatic events that were not work-related have you experienced/witnessed during COVID-19? | 4.5 (15.6) | 10.2 (46.2) | 7.3 (34.4)
Types of Work-Related Traumatic Events Experienced [Count of Participants; unit: Participants] — Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=42). Note, categories below are not mutually exclusive as participants may have experienced multiple categories of potentially traumatic events.
  Participants
    A traumatic or tragic death of a patient: number analyzed (Participants) | 42 | 42 | 84
    A traumatic or tragic death of a patient | 38 | 40 | 78
    A severe or unsuccessful resuscitation: number analyzed (Participants) | 42 | 42 | 84
    A severe or unsuccessful resuscitation | 26 | 32 | 58
    Witnessing events surrounding colleague who has fallen ill or died of COVID-19: number analyzed (Participants) | 42 | 42 | 84
    Witnessing events surrounding colleague who has fallen ill or died of COVID-19 | 19 | 18 | 37
    Situation where the care of a patient failed or did not go as planned: number analyzed (Participants) | 42 | 42 | 84
    Situation where the care of a patient failed or did not go as planned | 33 | 31 | 64
    Threats or violence against healthcare professionals: number analyzed (Participants) | 42 | 42 | 84
    Threats or violence against healthcare professionals | 26 | 13 | 39
    Event involving sudden increased risk of COVID-19 infection: number analyzed (Participants) | 42 | 42 | 84
    Event involving sudden increased risk of COVID-19 infection | 23 | 29 | 52
    A traumatic or tragic event where a patient reminded you of yourself, a family member or friend: number analyzed (Participants) | 42 | 42 | 84
    A traumatic or tragic event where a patient reminded you of yourself, a family member or friend | 29 | 31 | 60
    Event involving extremely distressed/grieving relatives of patients: number analyzed (Participants) | 42 | 42 | 84
    Event involving extremely distressed/grieving relatives of patients | 37 | 33 | 70
    Being faced with suicide / suicide attempt: number analyzed (Participants) | 42 | 42 | 84
    Being faced with suicide / suicide attempt | 14 | 18 | 32
    Other: number analyzed (Participants) | 42 | 42 | 84
    Other | 5 | 2 | 7
Timeframe of work-related traumatic events experienced at baseline [Count of Participants; unit: Participants] — Population: Please note, outcome options are not necessarily mutually exclusive.
  Participants
    Within the last 24 hours: number analyzed (Participants) | 42 | 42 | 84
    Within the last 24 hours | 3 | 4 | 7
    Within the past month: number analyzed (Participants) | 42 | 42 | 84
    Within the past month | 7 | 8 | 15
    Between 1-3 months ago: number analyzed (Participants) | 42 | 42 | 84
    Between 1-3 months ago | 8 | 7 | 15
    More than 3 months ago: number analyzed (Participants) | 42 | 42 | 84
    More than 3 months ago | 22 | 24 | 46
    Ongoing exposure to traumatic events is part of my job during the COVID-19 pandemic: number analyzed (Participants) | 42 | 42 | 84
    Ongoing exposure to traumatic events is part of my job during the COVID-19 pandemic | 33 | 37 | 70
Perceived threat to self/other [Mean (Standard Deviation); unit: units on a 10-point Likert scale] — Participants are asked to rate "to what extent did you feel your life was in danger?" and "to what extent did you think that someone else's life was in danger?" on a 10-point Likert scale from 0 (not at all) to 10 (extremely). This is based on the assessment of perceived life threat used in previous prospective studies following trauma (Blanchard et al., 1995), as used in Iyadurai et al. (2018). Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=41)
  units on a 10-point Likert scale
    Perceived life threat to someone else: number analyzed (Participants) | 41 | 42 | 83
    Perceived life threat to someone else | 9.1 (1.4) | 8.3 (2.8) | 8.7 (2.3)
    Perceived life threat to self: number analyzed (Participants) | 41 | 42 | 83
    Perceived life threat to self | 4.7 (3.4) | 5.3 (3.4) | 5.0 (3.4)
Peritraumatic Distress Inventory [Mean (Standard Deviation); unit: Total Score of Items] — This 13-item measure assesses the extent to which participants experienced a number of emotional reactions during the trauma (DSM-IV, criterion A2). Items are rated on a 5-point Likert scale from 0 (not at all) to 4 (extremely) and a total score is calculated as a sum of all 13-items (range 0-52). Higher scores indicate a higher level of distress. Population: Total n observed for data is 84 (delayed arm n=42; immediate arm n=41)
  Total Score of Items
    number analyzed (Participants) | 41 | 42 | 83
    (all) | 30.5 (10.2) | 28.6 (9.9) | 29.6 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Intrusive Memories of Traumatic Event(s)
Description: Number of intrusive memories of traumatic event(s) recorded by participants in a brief daily online diary for 7 days at week 4 (i.e., Day 22-28). To control for the number of intrusive memories recorded by participants in each experimental group during the run-in/screening week, we included the baseline count of intrusive memories (along with binary arm status) as fixed effect covariates in the Poisson regression model used for primary analysis.
Time Frame: Week 4
Population: All analyses were completed on an intention-to-treat basis as a between-group comparison.
Measure: Median (95% Confidence Interval); unit: Number of intrusive memories
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Number of intrusive memories
  Run-in/screening week | 14.5 [10.0 to 21.5] | 14.0 [8.0 to 19.0]
  Week 4 (Primary Outcome): number analyzed (Participants) | 36 | 39
  Week 4 (Primary Outcome) | 1.0 [0.0 to 3.0] | 10.0 [6.0 to 16.5]
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; For more information on analysis models see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — Poisson regression was performed with baseline measure and binary arm status included as fixed effect covariates. Various regression models for count data were compared to find the best fitting model. Visual exploratory data and model evaluation showed that the Zero Inflated Negative Binomial (ZINB) regression model provided the best fit and was used as the model for the ITT analysis of the primary outcome; p <= 0.001, Regression, Poisson — No multiplicity adjustments were applied as there was only one primary outcome, and secondary outcomes aimed to support the primary analyses. The a priori threshold for statistical significance was 0.05; Incidence Rate Ratio = 0.31, 95% CI 2-sided [0.20 to 0.48]; See also Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0

2. Secondary Outcome: Number of Intrusive Memories of Traumatic Event(s)
Description: Number of intrusive memories of traumatic event(s) recorded by participants in a brief daily online diary for 7 days.
  Total number of intrusive memories reported in Week 4 compared to run-in/screening week for the immediate intervention group and Week 8 compared to Week 4 for the delayed intervention group (i.e., within-group comparisons).
Time Frame: Run-in/screening week (immediate intervention arm), week 4 (both arms) and week 8 (delayed intervention arm)
Population: Analyses were completed on an intention-to-treat basis. After crossover, a within-subjects comparison pre-post intervention (week 4 - week 8) was completed for the comparator delayed intervention group. Please see participant flow.
Measure: Median (Inter-Quartile Range); unit: Number of intrusive memories
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Number of intrusive memories
  Run-in/screening week | 14.00 [8.0 to 19.0] | 14.50 [10.0 to 21.50]
  Week 4: number analyzed (Participants) | 39 | 36
  Week 4 | 10.00 [6.0 to 16.5] | 1.00 [0.0 to 3.0]
  Week 8 (Delayed Arm Only): number analyzed (Participants) | 32 | 0
  Week 8 (Delayed Arm Only) | 1.00 [0.0 to 2.50] |
Statistical Analysis 1: Comparison: Delayed Intervention Arm; Within the comparator arm, where participants had delayed access to the intervention (i.e., delayed arm crossover), the number of intrusive memories in week 8 was compared to week 4. For full information about statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — Single level general Poisson regression was used to quantify within arm changes of number of intrusive memories in the delayed intervention arm, comparing pre-intervention (week 4) to post-intervention (week 8); p <= 0.001, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; Single level general Poisson regression was used to quantify within arm changes of number of intrusive memories pre- to post-intervention; Incidence Rate Ratio = 0.31, 95% CI 2-sided [0.21 to 0.45]; For full results see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0
Statistical Analysis 2: Comparison: Immediate Intervention Arm; Within the immediate intervention arm, where participants had immediate access to the intervention, the number of intrusive memories in Week 4 was compared to the run-in/screening week. For full information about statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — Single level general Poisson regression was used to quantify within arm changes of number of intrusive memories in the immediate intervention arm, comparing pre-intervention (run-in/screening week) to post-intervention (week 4); p < 0.001, Regression, Poisson — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Incidence Rate Ratio = 0.22, 95% CI 2-sided [0.10 to 0.45]

3. Secondary Outcome: Intrusive Memory Ratings, Ordinal Items
Description: The 9-item questionnaire assesses a number of intrusive memories characteristics. These characteristics include frequency (7-point categorical response from 'never' to 'many times a day); distress (0=not at all to 10=extremely); disruption to concentration (0=not at all to 10=extremely); interference with what you were doing (how much (0=not at all to 10=extremely) and for how long (6-point categorical response from '<1min' to '+60mins')); impact on work functioning (0=not at all to 10=extremely) and in what ways (open text response)); impact on functioning in other areas of life (how much (0= not at all to 10 = extremely) and in what ways (open text response)).
  Five quantitative outcomes are presented here. For two further ordinal items, frequency and duration of interference, please see below.
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
score on a scale
  Baseline - How distressing were your intrusive memories?: number analyzed (Participants) | 43 | 42
  Baseline - How distressing were your intrusive memories? | 6.00 (1.83) | 6.02 (1.83)
  Week 4 - How distressing were your intrusive memories?: number analyzed (Participants) | 38 | 35
  Week 4 - How distressing were your intrusive memories? | 5.53 (1.94) | 2.86 (2.45)
  Week 8- How distressing were your intrusive memories? | 2.87 (2.67) | 2.00 (2.44)
  Baseline - How much did they disrupt your concentration?: number analyzed (Participants) | 43 | 42
  Baseline - How much did they disrupt your concentration? | 6.70 (1.88) | 7.05 (2.29)
  Week 4 - How much did they disrupt your concentration?: number analyzed (Participants) | 38 | 35
  Week 4 - How much did they disrupt your concentration? | 5.95 (1.72) | 2.74 (2.76)
  Week 8 - How much did they disrupt your concentration? | 2.67 (2.19) | 1.97 (2.40)
  Baseline - How much did they interfere with what you were doing?: number analyzed (Participants) | 43 | 42
  Baseline - How much did they interfere with what you were doing? | 5.42 (2.30) | 5.95 (2.26)
  Week 4 - How much did they interfere with what you were doing?: number analyzed (Participants) | 38 | 35
  Week 4 - How much did they interfere with what you were doing? | 5.13 (1.99) | 2.26 (2.32)
  Week 8 - How much did they interfere with what you were doing? | 2.27 (2.08) | 1.55 (2.01)
  Baseline - How much did your intrusive memories affect your work functioning?: number analyzed (Participants) | 43 | 42
  Baseline - How much did your intrusive memories affect your work functioning? | 4.53 (2.75) | 4.71 (2.64)
  Week 4 - How much did your intrusive memories affect your work functioning?: number analyzed (Participants) | 38 | 35
  Week 4 - How much did your intrusive memories affect your work functioning? | 3.97 (2.81) | 1.71 (2.63)
  Week 8 - How much did your intrusive memories affect your work functioning? | 1.93 (2.27) | 1.00 (1.65)
  Baseline - How much did your intrusive memories affect your functioning in other areas of your life?: number analyzed (Participants) | 43 | 42
  Baseline - How much did your intrusive memories affect your functioning in other areas of your life? | 5.30 (2.53) | 5.55 (2.21)
  Week 4 - How much did your intrusive memories affect your functioning in other areas of your life?: number analyzed (Participants) | 38 | 35
  Week 4 - How much did your intrusive memories affect your functioning in other areas of your life? | 4.42 (2.78) | 1.89 (2.35)
  Week 8 - How much did your intrusive memories affect your functioning in other areas of your life? | 1.53 (1.83) | 1.58 (2.57)
Statistical Analysis 1: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Intrusive memory ratings, 'How distressing were your intrusive memories?' (treatment effects for between-arm comparisons) at week 4. For full information on statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — Multilevel modelling (MLM) was performed with baseline measure, binary arm status, follow-up time and arm-by-time interaction included as fixed-effect covariates. Individual participant was also included as a level-two analytical unit, to quantify: (a) between-group treatment effect estimates and (b) within-group changes between each follow-up time for secondary outcome measures; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-3.72 to -1.54]; Please see Iyadurai et al., 2023 Supplementary Tables for within-subjects comparisons (Iyadurai, et al. Transl Psychiatry 13, 290 (2023). https://doi.org/10.1038/s41398-023-02578-0)
Statistical Analysis 2: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Intrusive memory ratings, 'How much did they disrupt your concentration?' (treatment effects for between-arm comparisons) at week 4. For full information on statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.21, 95% CI 2-sided [-4.28 to -2.15]; [other analysis details as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Intrusive memory ratings, 'How much did they interfere with what you were doing?' (treatment effects for between-arm comparisons) at week 4. For full information on statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-3.90 to -1.95]; Please see Iyadurai et al., 2023 Supplementary Tables for within-subjects comparisons. (Iyadurai, et al. Transl Psychiatry 13, 290 (2023). https://doi.org/10.1038/s41398-023-02578-0)
Statistical Analysis 4: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Intrusive memory ratings, 'How much did your intrusive memories affect your work functioning?' (treatment effects for between-arm comparisons) at week 4. For full information on statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-3.22 to -1.08]; [other analysis details as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Intrusive memory ratings, 'How much did your intrusive memories affect your functioning in other areas of your life?' (treatment effects for between-arm comparisons) at week 4. For full information on statistical analysis see Iyadurai et al 2023, https://doi.org/10.1038/s41398-023-02578-0; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-3.67 to -1.51]; [other analysis details as in outcome 3, analysis 3]

4. Secondary Outcome: Intrusive Memory Ratings, Frequency of Intrusive Memories Over Past Week
Description: The 9-item questionnaire assesses a number of intrusive memories characteristics. Five ordinal items are presented separately (see "Intrusive Memory Ratings, ordinal items"). Here we present one of the two categorical items. This item assesses the frequency of intrusive memories over the past week (7-point categorical response from 'never' to 'many times a day').
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis.
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Participants
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: number analyzed (Participants) | 43 | 42
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Never | 0 | 0
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Once | 0 | 1
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Twice | 1 | 0
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Every other day | 14 | 6
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Once a day | 7 | 6
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Several times a day | 18 | 28
  Baseline - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Many times a day | 3 | 1
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: number analyzed (Participants) | 38 | 35
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Never | 0 | 11
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Once | 1 | 6
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Twice | 2 | 5
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Every other day | 10 | 6
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Once a day | 7 | 4
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Several times a day | 15 | 2
  Week 4 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Many times a day | 3 | 1
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: number analyzed (Participants) | 30 | 31
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Never | 7 | 14
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Once | 12 | 3
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Twice | 3 | 7
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Every other day | 4 | 5
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Once a day | 1 | 0
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Several times a day | 2 | 2
  Week 8 - Approximately how often did intrusive memories of the traumatic event pop into your mind?: Many times a day | 1 | 0

5. Secondary Outcome: Intrusive Memory Ratings, Duration of Interference
Description: The 9-item questionnaire assesses a number of intrusive memories characteristics. Five ordinal items are presented separately (see "Intrusive Memory Ratings, ordinal items"). Here we present one of the two categorical items. This item assesses the duration for which an intrusive memory interfered with with what participants were doing (6-point categorical response from '<1min' to '+60mins').
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis.
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Participants
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: number analyzed (Participants) | 43 | 42
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: <1min | 17 | 16
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: 1-5mins | 21 | 17
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: 6-10mins | 3 | 9
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: 11-30mins | 1 | 0
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: 31-60mins | 1 | 0
  Baseline - Each time, for (approximately) how long did they interfere with what you were doing?: +60mins | 0 | 0
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: number analyzed (Participants) | 38 | 35
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: <1min | 15 | 27
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: 1-5mins | 19 | 8
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: 6-10mins | 3 | 0
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: 11-30mins | 1 | 0
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: 31-60mins | 0 | 0
  Week 4 - Each time, for (approximately) how long did they interfere with what you were doing?: +60mins | 0 | 0
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: number analyzed (Participants) | 30 | 31
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: <1min | 23 | 27
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: 1-5mins | 4 | 4
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: 6-10mins | 2 | 0
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: 11-30mins | 1 | 0
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: 31-60mins | 0 | 0
  Week 8 - Each time, for (approximately) how long did they interfere with what you were doing?: +60mins | 0 | 0

6. Secondary Outcome: Impact of Event Scale-Revised (IES-R)
Description: This 22-item questionnaire assesses subjective distress after a traumatic event (with reference to the events for which participants are taking part in the study).
  Items are rated for how distressing they have been during the past 7 days on a 5-point ordinal scale ranging from 0 ("not at all") to 4 ("extremely"). The measure consists of three subscales with subscale and total scores calculated as the mean of all items: intrusion subscale (8-items, score range 0-4), avoidance subscale (8-items, score range 0-4) and hyperarousal subscale (6-items, score range 0-4), and total score (all 22-items, score range 0-4). We will analyse total score as the mean of all 22-items, and subscales as the mean of items in each subscale separately. Higher scores indicate higher levels of subjective distress after a traumatic event.
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
score on a scale
  Baseline - Total Score: number analyzed (Participants) | 43 | 41
  Baseline - Total Score | 2.17 (0.71) | 2.24 (0.77)
  Week 4 - Total Score: number analyzed (Participants) | 38 | 32
  Week 4 - Total Score | 1.70 (0.56) | 0.83 (0.58)
  Week 8 - Total Score | 0.78 (0.66) | 0.58 (0.59)
  Baseline - Intrusion Subscale: number analyzed (Participants) | 43 | 41
  Baseline - Intrusion Subscale | 2.43 (0.80) | 2.52 (0.91)
  Week 4 - Intrusion Subscale: number analyzed (Participants) | 38 | 32
  Week 4 - Intrusion Subscale | 1.86 (0.67) | 0.87 (0.63)
  Week 8 - Intrusion Subscale | 0.85 (0.71) | 0.62 (0.62)
  Baseline - Avoidance Subscale: number analyzed (Participants) | 43 | 41
  Baseline - Avoidance Subscale | 2.22 (0.83) | 2.19 (0.81)
  Week 4 - Avoidance Subscale: number analyzed (Participants) | 38 | 32
  Week 4 - Avoidance Subscale | 1.95 (0.70) | 1.06 (0.75)
  Week 8 - Avoidance Subscale | 0.87 (0.83) | 0.68 (0.76)
  Baseline - Hyperarousal Subscale: number analyzed (Participants) | 43 | 41
  Baseline - Hyperarousal Subscale | 1.83 (0.93) | 2.03 (0.96)
  Week 4 - Hyperarousal Subscale: number analyzed (Participants) | 38 | 32
  Week 4 - Hyperarousal Subscale | 1.27 (0.68) | 0.53 (0.52)
  Week 8 - Hyperarousal Subscale | 0.60 (0.63) | 0.41 (0.55)
Statistical Analysis 1: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Impact of Event Scale-Revised Total Score (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.08 to -0.53]; Please see Iyadurai et al., 2023 Supplementary Materials for within-subjects comparisons. (Iyadurai, et al. Transl Psychiatry 13, 290 (2023). https://doi.org/10.1038/s41398-023-02578-0)
Statistical Analysis 2: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Impact of Event Scale-Revised Intrusion Subscale (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.27 to -0.62]; [other analysis details as in outcome 3, analysis 3]
Statistical Analysis 3: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Impact of Event Scale-Revised Avoidance Subscale (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.09 to -0.42]; [other analysis details as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Impact of Event Scale-Revised Hyperarousal Subscale (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-0.97 to -0.44]; [other analysis details as in outcome 3, analysis 3]

7. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5) 4-item Version
Description: This shortened 4-item version of the PCL-5 assesses symptoms of PTSD over the last month.
  Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total score ranges from 0 to 16 (cut-off for possible PTSD is 10 or above).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 4-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 4-item scale measure
  Baseline: number analyzed (Participants) | 42 | 43
  Baseline | 8.71 (3.64) | 8.0 (3.27)
  Week 4: number analyzed (Participants) | 31 | 38
  Week 4 | 4.26 (2.86) | 6.74 (2.62)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 2.35 (3.13) | 2.87 (2.53)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for PTSD Checklist for DSM-5 (PCL-5) 4-item version (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-3.52 to -1.07]; Please see Iyadurai et al., 2023 Supplementary Materials for within-subjects comparisons.(Iyadurai, et al. Transl Psychiatry 13, 290 (2023). https://doi.org/10.1038/s41398-023-02578-0)

8. Secondary Outcome: Sleep Condition Indicator (SCI)
Description: This 8-item scale measures sleep problems against the DSM-5 criteria for insomnia disorder.
  Item responses are each scored 0-4, with scores from 0 to 2 indicating threshold criteria for insomnia disorder. Total score ranges 0-32, with a higher score indicating better sleep (cut-off for possible insomnia disorder is a total score from 0 to 2).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 8-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 8-item scale measure
  Baseline: number analyzed (Participants) | 41 | 42
  Baseline | 12.37 (7.75) | 12.71 (6.62)
  Week 4: number analyzed (Participants) | 30 | 38
  Week 4 | 19.13 (8.27) | 12.71 (6.06)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 20.65 (7.75) | 19.23 (7.55)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for Sleep Condition Indicator (SCI) (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.38, 95% CI 2-sided [2.56 to 8.20]; [other analysis details as in outcome 6, analysis 1]

9. Secondary Outcome: Generalised Anxiety Disorder 2-item Scale (GAD-2)
Description: Items are rated for how often they have bothered the respondent over the last two weeks, from 0 ("not at all") to 3 ("nearly every day"). Total score is the sum of both items and ranges from 0 to 6 (cut-off for possible GAD is 3 or above).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 2-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 2-item scale measure
  Baseline: number analyzed (Participants) | 41 | 42
  Baseline | 3.83 (1.80) | 3.07 (1.81)
  Week 4: number analyzed (Participants) | 30 | 38
  Week 4 | 2.07 (1.91) | 2.84 (1.79)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 1.65 (1.98) | 1.29 (1.55)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for Generalised Anxiety Disorder 2-item scale (GAD-2) (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.05, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.68 to -0.17]; [other analysis details as in outcome 6, analysis 1]

10. Secondary Outcome: Patient Health Questionnaire 2-item Version (PHQ-2)
Description: This 2-item short-form self-report measure assesses symptoms of depression.
  Items are rated for how often they have bothered the respondent over the last two weeks, from 0 ("not at all") to 3 ("nearly every day"). Total score is the sum of both items and ranges from 0 to 6 (cut-off for possible major depressive disorder is 3 or above).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 2-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 2-item scale measure
  Baseline: number analyzed (Participants) | 41 | 42
  Baseline | 2.76 (1.48) | 2.26 (1.82)
  Week 4: number analyzed (Participants) | 30 | 38
  Week 4 | 1.53 (1.50) | 1.92 (1.62)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 1.23 (1.61) | 1.23 (1.87)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for Patient Health Questionnaire 2-item version (PHQ-2) (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p > .05, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.23 to 0.19]; [other analysis details as in outcome 7, analysis 1]

11. Secondary Outcome: Psychological Outcome Profiles (PSYCHLOPS)
Description: This measure consists of 4 questions that are scored and designed to assess the impact of a person's intrusive memories.
  Questions 1b, 2b, 3b, and 4 are scored. These have a six-point ordinal scale ranging from 0 to 5 and are summed to generate a total score from 0 to 20. Higher values indicate the person is more severely affected.
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 4-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 4-item scale measure
  Baseline: number analyzed (Participants) | 40 | 42
  Baseline | 14.20 (3.30) | 13.29 (2.94)
  Week 4: number analyzed (Participants) | 30 | 38
  Week 4 | 6.97 (4.78) | 12.13 (3.57)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 5.65 (4.29) | 6.03 (4.13)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for Psychological Outcome Profiles (PSYCHLOPS) (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.49, 95% CI 2-sided [-8.48 to -4.51]; [other analysis details as in outcome 6, analysis 1]

12. Secondary Outcome: World Health Organization Disability Assessment Schedule 12-item Version (WHODAS 2.0)
Description: The 12-item, self-report version of the WHODAS 2.0 will be used to assess difficulties in relation to the impact of intrusive memories.
  Respondents rate how much difficulty they have had in each area in the past 30 days, from 0 (none) to 4 (extreme or cannot do). The overall score is calculated as a percentage of the maximum possible score (i.e., 48 points).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 12-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 12-item scale measure
  Baseline: number analyzed (Participants) | 40 | 42
  Baseline | 25.0 (15.23) | 21.88 (14.96)
  Week 4: number analyzed (Participants) | 28 | 38
  Week 4 | 13.54 (11.94) | 22.37 (14.40)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 10.76 (10.65) | 11.90 (14.55)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for World Health Organization Disability Assessment Schedule 12-item version (WHODAS 2.0) (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.78, 95% CI 2-sided [-15.06 to -4.50]; [other analysis details as in outcome 6, analysis 1]

13. Secondary Outcome: 5-level European Quality of Life 5 Dimension (EQ-5D-5L)
Description: The 5-level version of the EuroQol-5D (EQ-5D-5L) is a brief measure for assessing general quality of life and health status.
  Items assess mobility, self-care, usual activities, pain/discomfort and anxiety/depression each on a 5-point scale. 5 items are scored on a 5-point ordinal scale from 'no problem' (1) to 'highest level of problems' (5). Respondents also self-rate their overall health today on a visual analogue scale from 0 (the worst health you can imagine) to 100 (the best health you can imagine). Scores are analysed separately (not summed).
  Here we present the 'overall health' visual analogue scale item.
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
units on a scale
  Baseline: number analyzed (Participants) | 40 | 42
  Baseline | 66.03 (19.40) | 67.83 (19.30)
  Week 4: number analyzed (Participants) | 28 | 38
  Week 4 | 78.68 (13.52) | 65.13 (21.51)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 76.29 (14.83) | 78.23 (18.17)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for 5-level European Quality of Life 5 Dimension (EQ-5D-5L) (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.01, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.32, 95% CI 2-sided [4.61 to 20.04]; Please see Iyadurai et al., 2023 for EQ-5D-5L subscale comparisons and Iyadurai et al., 2023 Supplementary Materials for within-subjects comparisons. (Iyadurai, et al. Transl Psychiatry 13, 290 (2023). https://doi.org/10.1038/s41398-023-02578-0)

14. Secondary Outcome: Scale of Work Engagement and Burnout (SWEBO)
Description: This 19-item self-report measure assesses work engagement and burnout. Respondents rate how often they have felt each descriptive item in the past two weeks, from 1 (not at all) to 4 (all the time).
  The work engagement subscale consists of 10-items assessing three dimensions (attentiveness, vigour, and dedication) with each dimension consisting of 4-, 3-, and 3-items respectively. Greater scores indicate a higher (i.e., better) degree of work engagement.
  The burnout subscale consists of 9-items assessing three dimensions (Engagement, Exhaustion, and Disengagement), with each dimension consisting of 3-items. Greater scores indicate a higher (i.e., functionally worse) degree of burnout.
  A mean score is calculated for the work engagement and burnout subscales, from individual items (for both subscales, scores range 1-4).
Time Frame: Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
score on a scale
  Baseline - Work Engagement Subscale: number analyzed (Participants) | 42 | 40
  Baseline - Work Engagement Subscale | 2.19 (0.53) | 2.03 (0.46)
  Week 4 - Work Engagement Subscale: number analyzed (Participants) | 38 | 28
  Week 4 - Work Engagement Subscale | 2.10 (0.48) | 2.59 (0.66)
  Week 8 - Work Engagement Subscale: number analyzed (Participants) | 31 | 31
  Week 8 - Work Engagement Subscale | 2.50 (0.62) | 2.66 (0.69)
  Baseline - Burnout Subscale: number analyzed (Participants) | 42 | 40
  Baseline - Burnout Subscale | 2.33 (0.50) | 2.45 (0.54)
  Week 4 - Burnout Subscale: number analyzed (Participants) | 38 | 28
  Week 4 - Burnout Subscale | 2.40 (0.61) | 1.80 (0.54)
  Week 8 - Burnout Subscale: number analyzed (Participants) | 31 | 31
  Week 8 - Burnout Subscale | 1.97 (0.61) | 1.82 (0.56)
Statistical Analysis 1: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Scale of Work Engagement and Burnout (SWEBO) - Work Engagement Subscale (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [0.20 to 0.71]; [other analysis details as in outcome 3, analysis 3]
Statistical Analysis 2: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for Scale of Work Engagement and Burnout (SWEBO) - Work Burnout Subscale (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p <= 0.001, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.87 to -0.34]; [other analysis details as in outcome 3, analysis 3]

15. Secondary Outcome: Sickness Absence
Description: Single item assessing self-reported number of sick days taken from work in the last 4 weeks. Total scoring includes total number of sick days.
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Number of sick days
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Number of sick days
  Baseline: number analyzed (Participants) | 40 | 42
  Baseline | 3.80 (6.91) | 3.21 (6.62)
  Week 4: number analyzed (Participants) | 28 | 38
  Week 4 | 3.79 (7.36) | 3.45 (7.61)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 1.42 (5.16) | 1.65 (5.47)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for Sickness absence (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p > .05, Regression, Multilevel Poisson — [p-value comment as in outcome 1, analysis 1]; Incidence Rate Ratio = 1.50, 95% CI 2-sided [0.64 to 3.51]; [other analysis details as in outcome 6, analysis 1]

16. Secondary Outcome: Intention to Leave Job
Description: This 3 items questionnaire is used to assess participants' intention to leave their job e.g. "I think a lot about leaving the job", each rated from 1 (strongly agree) to 5 (strongly disagree). The total score ranges 3 to 15, with a lower score indicating stronger intention to leave the job.
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Total score of 3-item scale measure
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 43 | 43
Total score of 3-item scale measure
  Baseline: number analyzed (Participants) | 40 | 42
  Baseline | 8.65 (3.79) | 9.19 (3.62)
  Week 4: number analyzed (Participants) | 28 | 38
  Week 4 | 9.36 (4.63) | 10.32 (3.35)
  Week 8: number analyzed (Participants) | 31 | 31
  Week 8 | 9.94 (4.62) | 10.26 (3.86)
Statistical Analysis 1: Comparison: Immediate Intervention Arm vs Delayed Intervention Arm; ITT analysis for Intention to leave job (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p > .05, Regression, Multilevel Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-2.20 to 0.49]; [other analysis details as in outcome 3, analysis 3]

17. Secondary Outcome: Weekly Work Pattern, Number of Days Worked
Description: One item asses the number of days worked in the last week (both with responses from 0 to 7 days).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Days worked
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Days worked
  Baseline - On how many days did you work this week?: number analyzed (Participants) | 43 | 42
  Baseline - On how many days did you work this week? | 3.14 (1.81) | 3.21 (1.80)
  Week 4 - On how many days did you work this week?: number analyzed (Participants) | 38 | 35
  Week 4 - On how many days did you work this week? | 3.26 (1.78) | 2.66 (2.13)
  Week 8 - On how many days did you work this week?: number analyzed (Participants) | 30 | 31
  Week 8 - On how many days did you work this week? | 2.83 (1.58) | 3.48 (1.84)
Statistical Analysis 1: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for number of days worked (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p > .05, Regression, Multilevel Poisson — [p-value comment as in outcome 1, analysis 1]; Incidence Rate Ratio = 0.80, 95% CI 2-sided [0.60 to 1.07]; [other analysis details as in outcome 6, analysis 1]

18. Secondary Outcome: Weekly Work Pattern, Number of Night Shifts Worked
Description: One item asses the number of night shifts worked in the last week (both with responses from 0 to 7).
Time Frame: Baseline, 4 weeks and 8 weeks
Population: Analyses were completed on an intention-to-treat basis.
Measure: Mean (Standard Deviation); unit: Nights worked
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Nights worked
  Baseline: number analyzed (Participants) | 43 | 42
  Baseline | 0.65 (1.07) | 1.0 (1.36)
  Week 4: number analyzed (Participants) | 38 | 35
  Week 4 | 0.55 (1.01) | 0.83 (1.25)
  Week 8: number analyzed (Participants) | 30 | 31
  Week 8 | 0.57 (0.97) | 0.77 (1.18)
Statistical Analysis 1: Comparison: Delayed Intervention Arm vs Immediate Intervention Arm; ITT analysis for number of nights worked (treatment effects for between-arm comparisons) at week 4; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < .05, Regression, Multilevel Poisson — [p-value comment as in outcome 1, analysis 1]; Incidence Rate Ratio = 1.09, 95% CI 2-sided [0.57 to 2.09]; [other analysis details as in outcome 6, analysis 1]

19. Other Pre Specified Outcome: Changes to Health and Work - Discrete Outcomes
Description: The 6-item questionnaire will be used to assess the occurrence of any new traumatic events (presented below); any additional stressful life events (e.g. relationship problems, financial problems), new treatments received, social support received, changes to the job, or changes to the number of hours worked per week since the last assessment (see Supplementary Table 4 in Iyadurai et al., 2023).
Time Frame: 4 weeks and 8 weeks (both arms)
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Participants
  Week 4 - Have you experienced or witnessed any new work-related traumatic events?: number analyzed (Participants) | 38 | 28
  Week 4 - Have you experienced or witnessed any new work-related traumatic events?: Yes | 19 | 11
  Week 4 - Have you experienced or witnessed any new work-related traumatic events?: No | 19 | 17
  Week 8 -Have you experienced or witnessed any new work-related traumatic events?: number analyzed (Participants) | 31 | 31
  Week 8 -Have you experienced or witnessed any new work-related traumatic events?: Yes | 9 | 16
  Week 8 -Have you experienced or witnessed any new work-related traumatic events?: No | 22 | 15

20. Other Pre Specified Outcome: Changes to Health and Work - Continuous Outcomes
Description: as for outcome 19
Time Frame: 4 weeks and 8 weeks (both arms)
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Mean (Standard Deviation); unit: Number of events experienced/witnessed
Arm/Group | Delayed Intervention Arm | Immediate Intervention Arm
Number analyzed (Participants) | 43 | 43
Number of events experienced/witnessed
  Week 4 - How many new work-related traumatic events have you experienced/witnessed?: number analyzed (Participants) | 38 | 28
  Week 4 - How many new work-related traumatic events have you experienced/witnessed? | 3.2 (6.7) | 1.6 (2.8)
  Week 8 - How many new work-related traumatic events have you experienced/witnessed?: number analyzed (Participants) | 31 | 31
  Week 8 - How many new work-related traumatic events have you experienced/witnessed? | 1.5 (3.8) | 2.3 (3.5)
  Week 4 - How many new traumatic events that were not work-related have you experienced/witnessed?: number analyzed (Participants) | 38 | 28
  Week 4 - How many new traumatic events that were not work-related have you experienced/witnessed? | 0.2 (0.6) | 0.1 (0.5)
  Week 8 - How many new traumatic events that were not work-related have you experienced/witnessed?: number analyzed (Participants) | 31 | 31
  Week 8 - How many new traumatic events that were not work-related have you experienced/witnessed? | 0.1 (0.3) | 0.4 (1.08)

21. Other Pre Specified Outcome: Support From Managers and From Family/Friends
Description: The 2 item questionnaire asks "During the COVID-19 pandemic, how well supported have you been by your supervisors/managers?" and "how well supported have you been by your family and friends?" The response is rated as "not at all", "quite a bit", "moderately", "quite a bit", or "extremely"
Time Frame: Baseline
Population: Analyses were completed on an intention-to-treat basis. Please see Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 41 | 42
Participants
  How well supported have you been by your supervisors/managers?: Not at all | 6 | 9
  How well supported have you been by your supervisors/managers?: A little bit | 15 | 14
  How well supported have you been by your supervisors/managers?: Moderately | 9 | 10
  How well supported have you been by your supervisors/managers?: Quite a bit | 7 | 7
  How well supported have you been by your supervisors/managers?: Extremely | 4 | 2
  How well supported have you been by your family & friends?: Not at all | 1 | 1
  How well supported have you been by your family & friends?: A little bit | 10 | 2
  How well supported have you been by your family & friends?: Moderately | 10 | 11
  How well supported have you been by your family & friends?: Quite a bit | 9 | 15
  How well supported have you been by your family & friends?: Extremely | 11 | 13

22. Other Pre Specified Outcome: Optimisation Assessment
Description: Rates of recruitment, intervention use/adherence, outcome measure completion and participant attrition will be assessed.
Time Frame: Baseline, 4 weeks and 8 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Feedback Questionnaire
Description: This measure assesses participants' feedback for the intervention. Eight quantitative items assess how easy, helpful, distressing, burdensome and acceptable participants found the intervention, how willing they would be to use it in the future, how confident they would be in recommending it to a friend and how much they feel it could be used to support staff within NHS ICUs, with each rated on a 11-point ordinal scale from 0 (not at all) to 10 (very).
  For all items, a higher score indicates greater acceptability for the intervention. The two items assessing distress and burden are reverse coded such that higher scores (e.g., 10) indicate lower distress and burden respectively.
  A total score of all eight ordinal items (range 0-80) is calculated as the sum of items.
Time Frame: Week 4 (immediate intervention arm), Week 8 (delayed intervention arm)
Measure: Mean (Standard Deviation); unit: Total summed score of 8-items
Arm/Group | Immediate Intervention Arm | Delayed Intervention Arm
Number analyzed (Participants) | 28 | 28
Total summed score of 8-items | 63.79 (11.54) | 65.14 (13.58)

24. Other Pre Specified Outcome: Optional Qualitative Interview
Description: Qualitative interview will consist of a number of questions designed to gain an in-depth understanding of participants' experience of using the intervention, including acceptability, improvement suggestions, training/psychoeducation materials, potential barriers/facilitators to recruitment and uptake, and support needed for remote intervention delivery.
Time Frame: Week 5 (immediate intervention arm), Week 9 (delayed intervention arm)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were surveyed throughout the trial from enrolment to 8-weeks.
Description: All participants were asked to report adverse events, including any additional stressful life events or regarding new treatments, with both passive (could be reported throughout the trial) and active surveillance (open ended questions at 4 and 8 weeks).
  All adverse events and serious adverse events were unrelated to the study intervention or procedures.
Groups:
- Received Digital Imagery-Competing Task Intervention: Brief digital imagery-competing task intervention: First session guided by a researcher. Included a memory cue followed by playing the brief digital imagery-competing task with mental rotation instructions.
  Thereafter, option to engage in self-administered/guided sessions after the first session and record their intrusive memories (symptom monitoring).
  Immediate arm participants received access to the brief digital imagery-competing task intervention plus symptom monitoring for 8 weeks. Delayed arm participants received access to the brief digital imagery-competing task intervention plus symptom monitoring for 4 weeks (after 4 weeks of usual care).
- Usual Care (i.e., Delayed Arm, Randomisation - Week 4): Delayed arm participants could continue to access usual care for 4 weeks from randomisation. After 4-weeks, participants then received access to the brief digital imagery-competing task intervention plus symptom monitoring for 4 weeks.
- Run-In Period: At baseline, participants completed a daily online intrusive memory diary for 7 days to record the number of intrusive memories to work-related traumatic events. Those who reported at least 3 intrusive memories during the baseline week were asked to complete questionnaires and were randomised. The total number of intrusive memories that each participant recorded was included as a baseline covariate in the statistical modelling.
Arm/Group | Received Digital Imagery-Competing Task Intervention | Usual Care (i.e., Delayed Arm, Randomisation - Week 4) | Run-In Period
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/43 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/43 | 0/102
Other Adverse Events (participants affected / at risk) | 4/78 | 2/43 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Digital Imagery-Competing Task Intervention (N=78) | Usual Care (i.e., Delayed Arm, Randomisation - Week 4) (N=43) | Run-In Period (N=102)
Chest infection with reduced foetal movement (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — Participant admitted to hospital: 'chest infection with reduced foetal movement'. No SAE or AE was related to the study intervention or procedures.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Digital Imagery-Competing Task Intervention (N=78) | Usual Care (i.e., Delayed Arm, Randomisation - Week 4) (N=43) | Run-In Period (N=102)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04992390/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04992390/SAP_001.pdf